CLINICAL TRIAL: NCT07076732
Title: Platelet Indices and WBCs to MPV Ratio in Correlation With Angiographic Profiling of Myocardial Infarction With Non-Obstructive Coronary Arteries (MINOCA) and Its Short-Term Outcomes
Brief Title: Platelet Indices and WBCs to MPV Ratio in Correlation With Angiographic Profiling of Myocardial Infarction With Non-Obstructive Coronary Arteries and Its Short-Term Outcomes
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Remon Saleh Adly, Lecturer of Cardiovascular, Faculty of Medicine, Sohag University, Sohag, Egypt., Sohag University
Other Study IDs: Soh-Med-25-1-1PD
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Platelet Indices; White Blood Cell; Mean Platelet Volume; Myocardial Infarction; Obstructive Coronary Arteries; Short-Term Outcomes
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Myocardial infarction with nonobstructive coronary arteries (MINOCA) patients
  Interventions: Other: Coronary Angiography; Other: SYNTAX Score
- Control group: Healthy control individual.
  Interventions: Other: Coronary Angiography; Other: SYNTAX Score

INTERVENTIONS:
Other: Coronary Angiography — Coronary angiograms will be acquired digitally for quantification.
Other: SYNTAX Score — Upon retrieval of a version from http://www.syntaxscore.com, the anatomical SYNTAX score will be implemented to numerically evaluate the intricacy of coronary lesions.

SUMMARY:
This study aims to evaluate the role of platelet indices and the [White blood cell (WBC) /mean platelet volume (MPV)] ratio in correlation with angiographic profiles of patients diagnosed with myocardial infarction with non-obstructive coronary arteries (MINOCA) to assess their predictive value for short-term clinical outcomes.

DETAILED DESCRIPTION:
Globally, ischemic heart disease remains a significant cause of death, and its prevalence constantly increases. Around 5-15% of acute myocardial infarction (AMI) patients show nonobstructive (<50% stenosis) coronary arteries, named myocardial infarction with nonobstructive coronary arteries (MINOCA).

There are two main phases of inflammation during myocardial infarction: the inflammatory phase and the proliferative phase. The white blood cell (WBC) count and its subtypes have been investigated as potential predictors of cardiovascular outcomes in patients with coronary artery disease (CAD), serving as inflammatory markers.

The mean platelet volume (MPV) is determined in the progenitor cell, the bone marrow megakaryocyte. The platelet volume is found to be associated with cytokines (thrombopoietin, interleukin-6, and interleukin-3) that regulate megakaryocyte ploidy and platelet number and result in the production of larger platelets.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both sexes.
* Patients with acute myocardial infarction (AMI). Myocardial infarction with nonobstructive coronary arteries (MINOCA) is diagnosed if a patient fulfilled the AMI criteria in the absence of obstructive coronary arteries (type I: <50% stenosis; or type II: no stenosis) as recommended by the recent American Heart Association statement that introduces an updated definition incorporating the 4th universal MI definition, which by agreement excludes Takotsubo syndrome and myocarditis from the eventual diagnosis of MINOCA.

Exclusion Criteria:

* Previous history of MI or coronary revascularization (PCI or bypass surgery) with acute/chronic infection.
* Autoimmune diseases.
* Systemic inflammatory disease.
* Patients on treatment therapy which critically affects inflammatory cell count.
* Patients with malignancy.
* Chronic kidney disease.
* Severe liver disease.
* Severe anemia.
* Fever (>38°C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This case-control study will be performed at Sohag University Hospitals after approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
White blood cell count to mean platelet volume ratio (WMR) | Within 6 hours of symptom onset
  White blood cell count to mean platelet volume ratio (WMR) will be recorded.

SECONDARY OUTCOMES:
Incidence of major adverse cardiovascular events | 1 month post-procedure
  Incidence of major adverse cardiovascular events (MACE) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.